CLINICAL TRIAL: NCT05614297
Title: Agreement Between Two Methods for Assessing Knee Joint Laxity in Patients With ACL Injuries
Brief Title: Agreement Between Rolimeter and Lachmeter in Patients With ACL Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Region MidtJylland Denmark (Other)
Responsible Party: Principal Investigator, Nanna Rolving, Senior researcher, Aarhus University Hospital
Other Study IDs: ACL agreement study 2022
Record Dates: First submitted 2022-11-03; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Anterior Cruciate Ligament Injuries; Laxity of Ligament
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Joint Instability

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with ACL injuries: Patients who have sustained an ACL injury, surgically or non-surgically treated.
  Interventions: Diagnostic Test: Knee joint laxity test

INTERVENTIONS:
Diagnostic Test: Knee joint laxity test — Patients seen in an outpatient clinic in connection with an ACL injury or in connection with short or long-term follow-up after ACL surgery, will undergo a clinical assessment of their knee injury as part of standard care. This includes an assessment of knee joint laxity using both the Rolimeter and the Lachmeter, to allow for an assessment of agreement between the two methods.
  Other Names: Rolimeter; Lachmeter

SUMMARY:
The study is a quality assurance study, aiming to determine the agreement between two different measurement instruments for assessing knee joint laxity in patients with ACL injuries.

The study aims to include 60 patients with previous ACL injury, recruited in an outpatient clinic at Aarhus University Hospital from September 2022 to March 2023. For patients who consent to participate in the study, their knee joint laxity in both the injured and the non-injured knee is assessed using both a Rolimeter and a Lachmeter. Subsequently, the collected data are examined to determined the agreement between the two measurement instruments.

DETAILED DESCRIPTION:
Methods:

In connection with their visit at either the orthopaedic or physiotherapy outpatient clinic, patients are invited to participate in the study. Patients consenting to participate will undergo knee joint laxity tests with both the Rolimeter and the Lachmeter, and in addition health-related and demographic data are collected.

The two tests are performed in random order for each patient, and the same physiotherapist conducts the two tests in each individual patient. The physiotherapist performing the two tests reads and notes the score on the first test, while a different physiotherapist, blinded to the score of the first test, reads and notes the score on the second test.

Agreement between the two scores are investigated using a Bland-Altman plot, with calculation of bias and upper and lower limits of agreements with 95% CIs. A priori, an acceptable difference between the two methods is set at 1 millimeter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ACL injury awaiting potential ACL-surgery
* Patients with previous ACL-surgery

Exclusion Criteria:

* Multiligament injury
* PCL injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are recruited consecutively from either the orthopaedic outpatient clinic (patients with ACL-injury) or the physiotherapy outpatient clinic (patients who have previously undergone ACL surgery) at Aarhus University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Knee joint laxity (millimeters) | For surgicaly treated patients: Between 1 year and up to 5 years post-surgery. For non-surgically treated patients: Up to 12 weeks after ACL injury.
  Measurement of knee joint laxity using both a Rolimeter and a Lachmeter is conducted in connection with the patients' visit at the outpatient clinic.

CONTACTS AND LOCATIONS:
Overall Officials: Nanna Rolving, PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No